CLINICAL TRIAL: NCT01590394
Title: Prospective Evaluation of Luminal Patency of a Prototype Large Plastic Biliary Stent in the Palliation of Malignant Distal Biliary Strictures.
Brief Title: Patency of a Prototype Large Plastic Biliary Stent in the Palliation of Malignant Distal Biliary Strictures.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling subjects and transporting scope for sterilization
Sponsor: Mayo Clinic (Other)
Collaborators: Olympus America, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher J. Gostout, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-003154
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Stricture; Obstruction; Cancer
Keywords: obstruction; bile duct; malignant
MeSH Terms: conditions — Constriction, Pathologic; Bites and Stings; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pancreatic Cancer Patients (Experimental): A large plastic biliary stent was placed in the bile duct.
  Interventions: Device: Large plastic biliary stent

INTERVENTIONS:
Device: Large plastic biliary stent — Stent placement for bile duct obstruction.

SUMMARY:
Plastic biliary stents which are a new larger size will remain free of obstructions for a longer period of time than currently used 10 French stents in cancer in the common bile duct.

DETAILED DESCRIPTION:
Malignant obstruction of the extra-hepatic bile duct often leads to jaundice and pruritus and occasionally results in cholangitis and bacteremia. Pancreatic cancer accounts for a large proportion of patients presenting with malignant extra-hepatic biliary obstruction. Most pancreatic cancers are unresectable at presentation, and palliation, including biliary decompression, is often a goal of therapy. Over the last decade, biliary decompression with endoscopically-placed stents during endoscopic retrograde cholangiopancreatography (ERCP) has largely replaced surgical bilioenteric diversion. Biliary decompression via endoscopic stenting alleviates cholestatic symptoms and improves quality of life. When compared to surgery, endoscopically placed plastic stents result in decreased morbidity and a trend towards decreased 30 day mortality. However, surgery is associated with a lower risk of recurrent biliary obstruction.

Stent diameter is an important factor in determining duration of biliary luminal patency. All plastic biliary stents will ultimately occlude due to deposition of bacterial biofilm. The original plastic biliary stents were 7 French (Fr) in diameter, with a patency rate of about 4 weeks. With increases in the size of the working channel of duodenoscopes, the limiting factor in what diameter stent can be deployed, 10 Fr stents were developed, with patency rates of approximately 15 weeks (3-4 months). Until recently, the largest stent that could be deployed with the current endoscopic technology using a conventional duodenoscope of acceptable outer diameter was 11.5 Fr; the limited available data suggest that these stents do not offer more prolonged luminal patency interval compared to 10 Fr stents.

In the early 1990s, self-expandable metal stents (SEMS) became available for use in palliation of malignant biliary obstruction. Once deployed, SEMS achieve larger diameters than plastic stents, which results in a longer median patency interval of approximately six to eight months.[3, 6, 9-12] Although effective, metal stents are eight to ten times more costly than plastic stents.

Recently, a large working channel duodenoscope with an acceptable outer diameter has been developed. This prototype duodenoscope allows passage of larger stents, which the investigators have successfully placed in select cases using this prototype. This duodenoscope, manufactured by Olympus Medical Systems Corp., is FDA approved.

The investigators hypothesize that, with the substantially increased luminal diameter, larger plastic stents will provide more prolonged relief of obstructive jaundice in patients with malignant distal common bile duct strictures. If this proves to be true, larger plastic stents may constitute a cost-effective alternative to SEMS, especially in health care systems that cannot afford SEMS.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. ≥ 18 and ≤ 85 years of age
2. Malignant biliary obstruction, known or suspected
3. Increased bilirubin or jaundice or history thereof
4. Duct stricture (obstruction) ≥ 1 cm distal to the biliary hilum (bifurcation of the common hepatic duct into the right and left hepatic ducts)
5. Not an operative candidate

Exclusion Criteria:

1. Unable to obtain consent
2. Unable to tolerate endoscopic procedure
3. Suspected non-malignant bile duct stricture
4. Candidate for potentially curative surgical intervention
5. Previous SEMS
6. Previous bile duct surgery
7. Diffuse liver metastasis
8. Peritoneal metastasis by CT
9. Presence of ascites
10. Duodenal obstruction preventing passage of the duodenoscope to the level of the papilla
11. Failure to cannulate bile duct during ERCP
12. Karnofsky performance score < 40

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Gostout, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at Mayo Clinic in Rochester, Minnesota.
Groups:
- Pancreatic Cancer Patients: A large plastic biliary stent was placed in the bile duct for bile duct obstruction.
Period: Overall Study
Arm/Group | Pancreatic Cancer Patients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pancreatic Cancer Patients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Large Plastic Biliary Stents Will Have a Longer Patency Time Than Conventionally Used 10 Fr Stents in Subjects as Compared to Well-known Published Historical Control Data.
Time Frame: 6 months
Population: Data were not analyzed, because there were too few subjects to make the outcome measure meaningful. Principal investigator retired before any analysis could be performed.
Arm/Group | Pancreatic Cancer Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pancreatic Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulty in enrolling subjects and transporting the scope for sterilization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes